CLINICAL TRIAL: NCT04707001
Title: Urinary Retention After Arthroplasty - UREA Trial
Brief Title: Urinary Retention After Arthroplasty
Acronym: UREA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1U/2020
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Urinary Retention Postoperative; Arthroplasty Complications

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound monitoring group (Active Comparator): In the ultrasound group, urinary retention is monitored, according to current practice, with an ultrasound scanner and the patient is catheterized if necessary, if residual urine exceeds 800 ml, or if the patient is symptomatic.
  Interventions: Other: Catheterization based on ultrasound
- Symptoms alone group (Active Comparator): Urination is monitored by asking at regular intervals about the onset of spontaneous urination and the patient is catheterized only on a symptomatic basis.
  Interventions: Other: Catheterization based on evaluation of symptoms

INTERVENTIONS:
Other: Catheterization based on ultrasound — Bladder volume ultrasound
  Arms: Ultrasound monitoring group
Other: Catheterization based on evaluation of symptoms — Ask for symptoms: Need to urinate, lower abdominal pain
  Arms: Symptoms alone group

SUMMARY:
Arthroplasty increases the risk of postoperative urinary retention. Treatment of postoperative urinary retention is indwelling or intermittent catheterization. The need for catheterization is most commonly determined with an ultrasound scanner. Catheterization increases the risk of urinary tract infection, which may further lead to haematogenic infection of the artificial joint. There is no evidence of an optimal way to monitor the onset of spontaneous urination.

The aim of the study is to determine whether monitoring the onset of spontaneous urination after fast track knee arthroplasty is safe based on symptoms alone without ultrasound monitoring.

DETAILED DESCRIPTION:
Adult patients undergoing knee arthroplasty will be recruited to this study. Participants will be randomized to the ultrasound monitoring group or the symptoms alone group. In the symptoms alone group, urination is monitored by asking at regular intervals about the onset of spontaneous urination and the patient is catheterized only on a symptomatic basis or if spontaneous voiding has not started 10 hours after the spinal anesthesia. Symptoms that indicate catheterization are lower abdominal pain or need to void. In the ultrasound group, urinary retention is monitored according to current practice with an ultrasound scanner and the patient is catheterized if residual urine exceeds 800 ml or if the patient is symptomatic.

The primary outcome variable is the change in IPSS score from the baseline to 3 months after the procedure. The baseline score is evaluated preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* elective total knee arthroplasty

Exclusion Criteria:

* previous surgery for urologic cancer
* fracture as indication for surgery
* lack of co-operation
* untreated urinary retention
* nephrostoma
* general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — in 1:1 ratio. Participant eligibility is based on self-representation of gender identity.
Enrollment: 170 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 3 months after surgery
  IPSS questionnaire compared to IPSS before surgery. The minimum score is 0. The maximum score is 35. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 12 months after surgery
  IPSS questionnaire compared to IPSS before surgery. The minimum score is 0. The maximum score is 35. Higher scores mean a worse outcome.
Incidence of urinary complications | 3 months after surgery
  Incidence of urinary complications
Health-related quality of life (15D) score | 3 months after surgery
  Health-related quality of life(15D) score compared to 15D score before surgery. The minimum score is 0. The maximum score is 1. Higher scores mean a better outcome.
Incidence of urinary complications | 12 months after surgery
  Incidence of urinary complications
Health-related quality of life (15D) score | 12 months after surgery
  Health-related quality of life(15D) score compared to 15D score before surgery. The minimum score is 0. The maximum score is 1. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Juha Paloneva, professor, Principal Investigator — Chief medical director; Heikki Seikkula, PhD, Study Chair — Investigator; Juho Sippola, MD, Study Chair — Investigator; Konsta Pamilo, PhD, Study Chair — Investigator; Jonne Åkerla, MD, Study Chair — Investigator; Aleksi Reito, PhD, Study Chair — Investigator; Pirkko Kinnunen, Study Chair — Investigator
Locations (1):
- Central Finland Hospital Nova, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No